CLINICAL TRIAL: NCT04842149
Title: The Effects of Bifidobacterium Breve Bif195 for Small Intestinal Crohn's Disease: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: The Effects of Bifidobacterium Breve Bif195 for Small Intestinal Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Chr Hansen A/S (Unknown)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Principal Investigator, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-20068527
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease
Keywords: Probiotics
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bif195 capsules (Active Comparator): The capsule will contain approximately 15*10^9 CFU of Bif195 per day. Excipients: Microcrystalline Cellulose 6 mg per capsule, Magnesium Stearate 1.5 mg per capsule, Maltodextrin 277.8 mg per capsule, and Sodium Ascorbate 14.7 mg per capsule.
  Interventions: Dietary Supplement: Bif195 capsules
- Placebo capsules (Placebo Comparator): The capsule contain only excipients: Microcrystalline Cellulose 6 mg per capsule, Magnesium Stearate 1.5 mg per capsule, Maltodextrin 277.8 mg per capsule, and Sodium Ascorbate 14.7 mg per capsule.
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Bif195 capsules — 1 capsule daily for 8 weeks
  Arms: Bif195 capsules
Dietary Supplement: Placebo capsules — 1 capsule daily for 8 weeks
  Arms: Placebo capsules

SUMMARY:
The purpose of this study is to investigate if the probiotic Bifidobacterium breve Bif195 (Bif195) will result in improvement in clinical outcome in patients with small intestinal Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory bowel disease (IBD) with an incidence rate at 11/100 000 per year in Denmark.

The disease can potentially affect the entire gastrointestinal tract, though the most common affected area is terminal ileum and the adjacent part of colon.

CD is a result of both genetic and environmental factors together with the intestinal microbiota, however the precise etiology is unclear.

A change of the intestinal microbiota with a reduced occurrence of e.g. Bacteroides species, Firmicutes and the anti-inflammatory bacteria Faecalibacterium prausnitzii is found in CD patients compared to healthy controls. Also a reduction of the mucosa-associated Bifidobacteria has been associated with the risk of mucosal inflammation.

The hypothesis that an imbalance between potentially beneficial and pathogenic bacteria contribute to the pathogenesis of IBD, including CD, has led to the suggestion that manipulation of the microbiota may be an attractive target for therapeutic interventions in IBD.

A new probiotic bacterium, Bifidobacterium breve Bif195 (Bif195) has been identified and has shown great effects on preventing enteropathy and ulcers on the gut mucosa in healthy volunteers given acetylsalicylic acid (13), and thereby Bif195 has also shown a potential in reducing gut permeability defects. This bacterium has not yet been investigated in CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with small intestinal CD
* Fecal calprotectin ≥ 250 ug/g
* IUS evidence of small bowel inflammation with wall thickness ≥ 4 mm
* At least 3 months af stable medical treatment
* Able to read and speak Danish

Exclusion Criteria:

* Positive rectal swab for pathogenic microorganisms
* Use of antibiotics, probiotics and systemic glucocorticosteroids within 4 weeks prior to inclusion
* Participation in other clinical trials within 30 days prior to inclusion
* Pregnancy, planned pregnancy or breast feeding
* Psychiatric disease
* Abuse of alcohol or drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Bowel Wall Thickness (BWT) from baseline measured by intestinal ultrasound (IUS) at 8 weeks | 8 weeks
  IUS will be performed in the non-fasting patient lying in supine position with a high-end ultrasound machine (Siemens Sequoia) with 10L4 transducer.

SECONDARY OUTCOMES:
Change in fecal calprotectin level from baseline at 8 weeks | 8 weeks
  measured from a fecal sample
Change in severity of symptoms from baseline measured by Harvey-Bradshaw index (HBI) at 8 weeks | 8 weeks
  HBI is a disease activity index for Crohns disease and consists of clinical parameters
Change in quality of life from baseline measured by Inflammatory Bowel Disease Questionnaire (IBDQ) Questionnaire Scores at 8 weeks | 8 weeks
  The IBDQ is a widely used instrument to assess QoL among IBD patients and consists of 32 questionaire
The change from baseline on Color Doppler Imaging Score (0-3) including inflammatory fat and ulceration (yes/no) at 8 weeks | 8 weeks
  measured by intestinal ultrasound (IUS)
Adverse and severe adverse events | 16 weeks
  Registered, if any events. Reported according to IHC-GCP

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD, PhD, Principal Investigator — Gastrounit, Copenhagen University Hospital Hvidovre, Copenhagen
Locations (1):
- Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gronbaek IMB, Halkjaer SI, Mollerup S, Hansen EH, Paulsen SJ, Engel S, Theede K, Wilkens R, Boysen T, Petersen AM. The effects of probiotic treatment with Bifidobacterium breve, Bif195 for small intestinal Crohn's disease and the gut microbiome: results from a randomised, double-blind, placebo-controlled trial. Gut Pathog. 2025 Apr 9;17(1):19. doi: 10.1186/s13099-025-00692-6. PMID 40205497